CLINICAL TRIAL: NCT03354767
Title: Observational Study Into the Effect on Muscle Wasting and Multiple Organ Function of Ischaemia-reperfusion Injury After Major Aortic Surgery
Brief Title: The Role of Ischaemia-reperfusion Injury in the Pathogenesis of Muscle Wasting After Thoracic Aortic Surgery
Acronym: RIMMAS
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: ImperialC
Record Dates: First submitted 2016-11-11; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2013-04

CONDITIONS: Muscular Diseases
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Plasma
  2. Serum
  3. Whole blood
  4. Skeletal muscle

GROUPS / COHORTS (2):
- Wasting patients: Patients with >10% loss of skeletal muscle one week after major aortic surgery
  Interventions: Procedure: Aortic and aortic valve surgery
- Non-wasting patients: Patients with <10% loss of skeletal muscle one week after major aortic surgery
  Interventions: Procedure: Aortic and aortic valve surgery

INTERVENTIONS:
Procedure: Aortic and aortic valve surgery

SUMMARY:
Single-centre observational study over one year investigating the mechanisms of muscle homeostasis in patients with acute skeletal muscle atrophy following major aortic surgery

DETAILED DESCRIPTION:
Some patients who are critically ill develop a syndrome of muscle weakness called Intensive Care Unit Acquired Paresis. This syndrome involves the development of severe muscle wasting and weakness and affects all skeletal muscles including the muscles which help one breathe. Muscle wasting and weakness whilst critically ill cause prolongation of mechanical ventilation, longer stays on the ICU, reduced mobility and prolonged rehabilitation in survivors. It has also been shown to increase the risk of death on ICU, due to an inability to wean patients from mechanical ventilation. Most patients recover; however in some, the effects last for many years and patients may not recover fully.

Although there is some understanding of why this syndrome develops, the molecular processes underlying the muscle wasting are not well understood. From the current scientific evidence, the investigators have identified a group or family of proteins believed to be important in the development of this condition, the activity of which are regulated by disease processes thought to lead to Intensive Care Unit Acquired Paresis (e.g. infection, inflammation, oxidative stress, immobility).

This research aims to investigate the role of these proteins in human tissue from patients who are at risk of Intensive Care Unit Acquired paresis. Even patients who do not go on to develop the full syndrome, in the early stages of ICU care, show some signs of muscle changes and loss of strength.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18) patients undergoing major aortic or aortic valve surgery

Exclusion Criteria:

* Pre-existing cause for neuromuscular weakness or severe wasting (such as previous stroke, neuromuscular disease or malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing major aortic or aortic valve surgery requiring cardiopulmonary bypass and aortic cross-clamping
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Rectus Femoris muscle cross-sectional area (%) | 7 days
  Percentage change in cross sectional area of Rectus Femoris muscle (cm2) in the first post-operative week, from pre-operative measurement (measured the day before surgery), repeated on day 7 post-operatively

IPD SHARING:
Plan to Share IPD: No